CLINICAL TRIAL: NCT01253694
Title: Ranibizumab in Residual Diabetic Macular Edema Following Previous Intravitreal Bevacizumab Therapy
Brief Title: Ranibizumab as a Rescue Therapy for Diabetic Macular Edema
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: New England Retina Associates (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DME-NERA
Record Dates: First submitted 2010-11-30; First posted 2010-12-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetes; edema; ranibizumab; bevacizumab; refractory
MeSH Terms: conditions — Diabetes Mellitus; Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with 3-5 consecutive Avastin injections (Experimental): These patients will receive 0.5 mg of intravitreal Ranibizumab monthly for 6 months.
  Interventions: Drug: injection of 0.5 mg of Intravitreal Ranibizumab
- Patients with 6 or more consecutive injections of Bevacizumab (Experimental): Patients will receive 0.5 mg of intravitreal Ranibizumab during the first 6 months.
  Interventions: Drug: injection of 0.5 mg of Intravitreal Ranibizumab

INTERVENTIONS:
Drug: injection of 0.5 mg of Intravitreal Ranibizumab — Following the sterile technique, intravitreal injection of anti-VEGF is applied
  Other Names: Lucentis

SUMMARY:
Treatment with Ranibizumab of the residual diabetic edema in patients with failed response to Bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible if the following criteria are met:

1. Age > 18 years
2. Diagnosis of diabetes mellitus (type 1 or 2)
3. Residual edema as determined by mean foveal thickness on Spectralis OCT (optical coherence tomography) > 300 microns and leakage seen on FA at baseline
4. Clinical evidence of retinal thickening due to macular edema involving the center of the macula, associated with diabetic retinopathy.
5. Previous history of at least 3-5 or more consecutive 1.25 mg of intravitreal bevacizumab injections for the treatment of diabetic macular edema (consecutive injections administered no more than 6 weeks apart).
6. BCVA of 20/32-20/400 using Early Treatment Diabetic Retinopathy Study (ETDRS)
7. Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography

Exclusion Criteria:

1. Pregnancy (positive pregnancy test) or known to be pregnant; also pre-menopausal women not using adequate contraception.
2. Participation in another ocular investigation or trial simultaneously.
3. Systemic use of anti-VEGF within 3 months prior to day 0.
4. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110)
5. Any condition that, in the opinion of the investigator, would preclude participation in the study (e.g. chronic alcoholism, drug abuse).
6. Evidence of vitreoretinal interface abnormality after ocular exam or OCT that may be contributing to the macular edema.
7. An eye that, in the investigator's opinion, has no chance of improving in visual acuity following resolution of macular edema (e.g. presence of subretinal fibrosis, ischemic maculopathy or geographic atrophy).
8. Presence of another ocular condition that may affect the visual acuity or macular edema during the course of the study (e.g. Age-related Macular Degeneration, uveitis, Irvine-Gass).
9. Evidence of active neovascularization of the iris or retina.
10. Evidence of central atrophy or fibrosis in the study eye.
11. Presence of substantial cataract, one that might decrease the vision by 3 or more lines of vision at sometime during the study.
12. History of vitreous surgery in the study eye.
13. History of cataract surgery within 6 months of enrollment.
14. History of YAG capsulotomy within 2 months of enrollment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with resolution of diabetic macular edema compared to baseline as determined by mean foveal thickness on Spectralis < 300 microns. | 6 months

SECONDARY OUTCOMES:
Evaluate the main change in BCVA (best corrected visual acuity) score over time | 6-12 months
  They will evaluate the amount of patients gaining 3 or more letters and the amount of patients losing 3 or more letters.

CONTACTS AND LOCATIONS:
Overall Officials: Nauman Chaudhry, MD, Principal Investigator — New England Retina Associates
Locations (1):
- New England Retina Associates, Norwich, Connecticut, United States